CLINICAL TRIAL: NCT00540449
Title: A Phase III, Randomized, Double-blind Trial of TMC278 25 mg q.d. Versus Efavirenz 600mg q.d. in Combination With a Fixed Background Regimen Consisting of Tenofovir Disoproxil Fumarate and Emtricitabine in Antiretroviral-naive HIV-1 Infected Subjects.
Brief Title: TMC278-TiDP6-C209: A Clinical Trial in Treatment Naive HIV-1 Patients Comparing TMC278 to Efavirenz in Combination With Tenofovir + Emtricitabine.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Tibotec Pharmaceuticals, Ireland (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CR002689; TMC278-TIDP6-C209 (Other: Tibotec Pharmaceuticals, Ireland); NCT00613639 (obsolete NCT alias)
Record Dates: First submitted 2007-10-04; First posted 2007-10-08 (Estimated); Results first posted 2011-07-11 (Estimated); Last update posted 2016-03-29 (Estimated); Status verified 2016-02

CONDITIONS: HIV Infections; HIV-1; Human Immunodeficiency Virus Type 1
Keywords: TMC278-C209; Antiretroviral; Non-nucleoside reverse transcriptase inhibitor; HIV-1; AIDS; TMC278-TiDP6-C209; Treatment Naive
MeSH Terms: conditions — HIV Infections; Acquired Immunodeficiency Syndrome | interventions — Rilpivirine; efavirenz

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Efavirenz (Active Comparator): Efavirenz 600mg once daily for 96 weeks
  Interventions: Drug: Efavirenz
- TMC278 (Experimental): TMC278 25 mg tablet once daily for 96 weeks
  Interventions: Drug: TMC278

INTERVENTIONS:
Drug: TMC278 — 25 mg tablet once daily for 96 weeks
  Arms: TMC278
Drug: Efavirenz — 600mg once daily for 96 weeks
  Arms: Efavirenz

SUMMARY:
The purpose of this trial is to compare the effectiveness, safety and tolerability of TMC278 given at a dose of 25 mg once daily versus efavirenz (EFV) at a dose of 600 mg once daily, when combined with a fixed background regimen consisting of emtricitabine (FTC) + tenofovir disoproxil fumarate (TDF), in HIV-1 infected patients who have not yet taken any anti-HIV drugs. The following evaluations will be done: antiviral activity, immunologic changes, and viral geno-/phenotype evolution, relationship of Pharmacokinetics (PK) and PK/Pharmacodynamics, medical resource utilization and treatment adherence.

DETAILED DESCRIPTION:
Over the past decade, anti-human immunodeficiency virus (HIV) drugs have been introduced sequentially for use in the clinic. Currently, patients are routinely being treated with 3 or 4 drug combinations including nucleoside/tide analogue reverse transcriptase inhibitors (NRTIs/NtRTIs), non-nucleoside reverse transcriptase inhibitors (NNRTIs), protease inhibitors (PIs), and/or fusion inhibitors. New potent antiretroviral (ARV) compounds that work in people whose HIV-1 virus is resistant to available drugs are urgently needed. This is a Phase III, randomized (study medication is assigned by chance), double-blind (neither the study physician nor the patient knows the name of the study assigned medication), double-dummy, active-controlled trial to compare the effectiveness, safety, and ability to tolerate TMC278 versus efavirenz (EFV). The study will last for 104 weeks which includes a screening period of 4 weeks, a 96-week treatment period, followed by a 4 week follow-up period. Patients will be randomly assigned to TMC278 or to efavirenz, either of these treatments will be in combination with two other anti-HIV drugs (2 NRTIs: emtricitabine (FTC) + tenofovir (TDF)). TDF/FTC will be administered as a fixed dose combination if available. The hypothesis to be provided in this study is that the investigational drug TMC278 will perform just like efavirenz (EFV) in terms of antiviral effectiveness (i.e., suppressing of the plasma viral load to a level < 50 HIV-1 RNA (ribonucleic acid) copies/mL) in ARV-naïve HIV-infected patients. During the trial, patients' health will be monitored by physical examination, interview to assess health and well being, and laboratory testing on blood and urine samples. Experimental Group: One tablet of TMC278 25 mg once daily plus one tablet of placebo once daily that looks just like efavirenz (EFV) plus tenofovir/emtricitabine; Control Group: One tablet of Placebo once daily that looks just like TMC278 plus EFV 600 mg once daily plus tenofovir/emtricitabine.

ELIGIBILITY:
Inclusion Criteria:

* Patient with documented HIV-1 infection
* Patient has never been treated with a therapeutic HIV vaccine or an ARV drug prior to screening
* Patient's HIV-1 plasma viral load at screening is > 5,000 HIV-1 RNA copies/mL (assayed by RNA PCR standard specimen procedure)
* Patient's virus is sensitive to TDF and FTC
* Patient agrees not to start ART (antiretroviral treatment) before the baseline visit

Exclusion Criteria:

* Previous use of ANY ARV drug for ANY length of time
* Any documented evidence of NNRTI resistance associated mutations in patient's HIV
* Category C AIDS defining illness, except: stable Kaposi Sarcoma, wasting syndrome if not progressive
* Pneumocystis carinii pneumonia (PCP) that is considered not cured
* Active TB
* Allergy or hypersensitivity to study or background ARTs
* Specific grade 3 or 4 toxicity
* Kidney impairment: calculated creatinine clearance <50 ml/min

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 694 (Actual)
Dates: Start 2008-05; Primary Completion 2010-02 (Actual); Study Completion 2011-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tibotec Pharmaceuticals Clinical Trial, Study Director — Tibotec Pharmaceutical Limited
Locations (92):
- United States (32):
  - Birmingham, Alabama
  - Phoenix, Arizona
  - Beverly Hills, California
  - Los Angeles, California
  - Newport Beach, California
  - Sacramento, California
  - Washington D.C., District of Columbia
  - Fort Lauderdale, Florida
  - Miami, Florida
  - Tampa, Florida
  - Vero Beach, Florida
  - West Palm Beach, Florida
  - Macon, Georgia
  - Chicago, Illinois
  - Baltimore, Maryland
  - Newark, New Jersey
  - Albany, New York
  - Buffalo, New York
  - New York, New York
  - Chapel Hill, North Carolina
  - Durham, North Carolina
  - Winston-Salem, North Carolina
  - Akron, Ohio
  - Cincinnati, Ohio
  - Columbus, Ohio
  - Portland, Oregon
  - Philadelphia, Pennsylvania
  - Columbia, South Carolina
  - Austin, Texas
  - Dallas, Texas
  - Seattle, Washington
  - Milwaukee, Wisconsin
- Argentina (3):
  - Buenos Aires
  - Córdoba
  - Guernica
- Australia (4):
  - Darlinghurst
  - Melbourne
  - Perth
  - Surry Hills
- Austria (2):
  - Innsbruck
  - Vienna
- Brazil (5):
  - Curitiba
  - Nova Iguaçu
  - Rio de Janeiro
  - Salvador
  - São Paulo
- Canada (3):
  - Ottawa, Ontario
  - Toronto, Ontario
  - Montreal, Quebec
- Denmark (3):
  - Copenhagen
  - Hvidovre
  - Odense
- France (5):
  - Loiré
  - Lyon
  - Paris
  - Tourcoing
  - Villejuif
- Mexico (2):
  - Mexico City
  - Zapopan
- Rotterdam, Netherlands
- Portugal (4):
  - Amadora
  - Lisbon
  - Portimão
  - Porto
- San Juan, Puerto Rico
- Romania (3):
  - Bucharest
  - Iași
  - Timișoara
- Russia (2):
  - Krasnodar
  - Saint Petersburg
- South Africa (6):
  - Bloemfontein
  - Cape Town
  - Durban
  - Houghton, Johannesburg
  - Johannesburg
  - Pretoria
- Spain (3):
  - Alicante
  - Barcelona
  - Madrid
- Sweden (3):
  - Gothenburg
  - Malmo
  - Stockholm
- Taiwan (4):
  - Kaohsiung City
  - Kaohsiung County
  - Tainan
  - Taipei
- Thailand (3):
  - Bangkok
  - Chiang Mai
  - Khon Kaen
- United Kingdom (3):
  - Birmingham
  - Brighton
  - London

REFERENCES:
- [Derived] Rimsky L, Van Eygen V, Hoogstoel A, Stevens M, Boven K, Picchio G, Vingerhoets J. 96-Week resistance analyses of rilpivirine in treatment-naive, HIV-1-infected adults from the ECHO and THRIVE Phase III trials. Antivir Ther. 2013;18(8):967-77. doi: 10.3851/IMP2636. Epub 2013 May 28. PMID 23714781
- [Derived] Nelson M, Amaya G, Clumeck N, Arns da Cunha C, Jayaweera D, Junod P, Li T, Tebas P, Stevens M, Buelens A, Vanveggel S, Boven K; ECHO and THRIVE Study Groups. Efficacy and safety of rilpivirine in treatment-naive, HIV-1-infected patients with hepatitis B virus/hepatitis C virus coinfection enrolled in the Phase III randomized, double-blind ECHO and THRIVE trials. J Antimicrob Chemother. 2012 Aug;67(8):2020-8. doi: 10.1093/jac/dks130. Epub 2012 Apr 24. PMID 22532465
- [Derived] Molina JM, Cahn P, Grinsztejn B, Lazzarin A, Mills A, Saag M, Supparatpinyo K, Walmsley S, Crauwels H, Rimsky LT, Vanveggel S, Boven K; ECHO study group. Rilpivirine versus efavirenz with tenofovir and emtricitabine in treatment-naive adults infected with HIV-1 (ECHO): a phase 3 randomised double-blind active-controlled trial. Lancet. 2011 Jul 16;378(9787):238-46. doi: 10.1016/S0140-6736(11)60936-7. PMID 21763936

RESULTS

PARTICIPANT FLOW:
Recruitment Details: One hundred and twelve sites in 21 countries randomized participants. In total, 694 participants were randomized: four participants did not start treatment and 690 participants started treatment (346 in the TMC278 group and 344 in the efavirenz [control ] group).
Groups:
- TMC278: 25 milligram (mg) tablet once daily for 96 weeks.
- Efavirenz: 600 mg once daily for 96 weeks.
Period: Overall Study
Arm/Group | TMC278 | Efavirenz
Started | 346 | 344
Completed | 262 | 266
Not Completed | 84 | 78
Not completed — Adverse Event | 12 | 32
Not completed — Sponsor's Decision | 1 | 1
Not completed — Subject Ineligible To Continue The Trial | 2 | 1
Not completed — Lost to Follow-up | 19 | 17
Not completed — Subject Non-Compliant | 7 | 5
Not completed — Subject Reached A Virologic Endpoint | 32 | 8
Not completed — Withdrawal by Subject | 10 | 10
Not completed — Other | 1 | 4

BASELINE CHARACTERISTICS:
Population: The analysis population included intent to treat (ITT) population defined as all randomized participants who received at least one dose of the study medication.
Groups:
- Total: Total of all reporting groups
Arm/Group | TMC278 | Efavirenz | Total
Number analyzed (Participants) | 346 | 344 | 690
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 1 | 0 | 1
  Between 18 and 65 years | 343 | 343 | 686
  >=65 years | 2 | 1 | 3
Age, Continuous [Mean (Standard Deviation); unit: years] | 37 (9.68) | 36.7 (9.51) | 36.8 (9.59)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 78 | 69 | 147
  Male | 268 | 275 | 543
Region Enroll [Number; unit: participants]
  Africa | 32 | 31 | 63
  Asia | 47 | 51 | 98
  Latin America | 60 | 69 | 129
  USA, Canada, Europe, Australia | 207 | 193 | 400

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Virological Response (Intent-to-Treat - Time to Loss of Virologic Response [TLOVR], <50 Copies/ml) at Week 48
Description: Virological response is defined as confirmed plasma viral load less than (<) 50 human immunodeficiency virus-1 (HIV-1) (ribonucleic acid [RNA]) copies/milliliter (ml) at Week 48. The TLOVR algorithm was used to derive response. Response needed to be confirmed at 2 consecutive visits and participants who permanently discontinued were considered nonresponders after discontinuation. Resuppression after confirmed virologic failure was considered as failure. Virologic Failure includes participants who were rebounder (confirmed viral load >= 50 copies/ml after being responder) or who were never suppressed (no confirmed viral load <50 copies/ml).
Time Frame: Week 48
Population: The ITT analysis set was considered the primary efficacy analysis set.
Measure: Number; unit: Participants
Arm/Group | TMC278 | Efavirenz
Number analyzed (Participants) | 346 | 344
Participants
  Responder | 287 | 285
  Virologic failure | 38 | 15
  Discontinued due to Adverse Event (AE) | 6 | 25
  Discontinued due to other reason than AE | 15 | 19
Statistical Analysis 1: Comparison: TMC278 vs Efavirenz; Assuming a response rate of 75% at 48 weeks for both treatment groups, 340 subjects were needed per treatment (TMC278 or EFV) to establish non-inferiority of TMC278 versus EFV with a maximum allowable difference of 12% and a 1-sided significance level of 2.5%, to yield 95% power; Test type: Non-Inferiority or Equivalence — If the lower limit of the 95% 2-sided confidence interval of the difference in proportions (TMC278 - EFV) exceeds -12%, non-inferiority of TMC278 versus EFV can be concluded; p < 0.0001, Regression, Logistic — Significance level was set at 2.5% (one-sided). No adjustment of p-value for multiple comparisons, since there was only single comparison for the primary endpoint; Logistic regression model included treatment arm as factor and baseline (log10) viral load as covariate; Difference in proportion of response = -0.4, 95% CI [-5.9 to 5.2] — Difference in proportion responders was estimated through the logistic regression model

2. Secondary Outcome: The Number of Participants With Virological Response (Intent-to-Treat - Snapshot, <50 Copies/ml) at Week 48
Description: The analysis is based on the last observed viral load (VL) data within the Week 48 window. Virologic response is defined as a VL<50 copies/ml (observed case). Missing VL was considered as non-response. Virologic Failure includes subjects who had VL>=50 copies/ml in the Wk48 window, subjects who discontinued early due to lack or loss of efficacy, subjects who discontinued for reasons other than an adverse event, death or lack or loss of efficacy and at the time of discontinuation had a VL>=50 copies/ml and subjects who had a switch in background regimen that was not permitted by the protocol.
Time Frame: Week 48
Population: The ITT analysis set was considered the primary efficacy analysis set.
Measure: Number; unit: Participants
Arm/Group | TMC278 | Efavirenz
Number analyzed (Participants) | 346 | 344
Participants
  Virologic Response HIV RNA <50 copies/mL at Wk 48 | 285 | 281
  Virologic Failure | 47 | 24
  No Viral Load Data in 48 week window | 14 | 39
Statistical Analysis 1: Comparison: TMC278 vs Efavirenz; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; p < 0.0001, Regression, Logistic; Logistic regression model included treatment arm as factor and baseline (log10) viral load as covariate; Difference in proportion of response = 0.3, 95% CI [-5.4 to 5.9] — Difference in proportion responders was estimated through the logistic regression model

3. Secondary Outcome: Number of Participants With Virological Response (Intent-to-Treat - Time to Loss of Virologic Response [TLOVR], <50 Copies/ml) at Week 96
Time Frame: Week 96
Population: The ITT analysis set was considered the primary efficacy analysis set.
Measure: Number; unit: Participants
Arm/Group | TMC278 | Efavirenz
Number analyzed (Participants) | 346 | 344
Participants
  Responder | 263 | 271
  Virologic failure | 45 | 16
  Death | 0 | 3
  Discontinued due to AE | 10 | 29
  Discontinued due to other reason than AE | 28 | 25
Statistical Analysis 1: Comparison: TMC278 vs Efavirenz; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.0055, Regression, Logistic; Logistic regression model included treatment arm as factor and baseline (log10) viral load as covariate; Difference in proportion of response = -3.2, 95% CI [-9.4 to 3.1] — Difference in proportion responders was estimated through the logistic regression model

4. Secondary Outcome: The Number of Participants With Virological Response (Intent-to-Treat - Snapshot, <50 Copies/ml) at Week 96
Time Frame: Week 96
Population: The Intent-to-Treat analysis set was considered the primary efficacy analysis set.
Measure: Number; unit: Participants
Arm/Group | TMC278 | Efavirenz
Number analyzed (Participants) | 346 | 344
Participants
  Virologic Response, <50 copies/ml | 265 | 268
  Virologic failure | 54 | 27
  No viral load data in the 96 week window | 27 | 49
Statistical Analysis 1: Comparison: TMC278 vs Efavirenz; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.0013, Regression, Logistic; Logistic regression model included treatment arm as factor and baseline (log10) viral load as covariate; Difference in proportion of response = -1.7, 95% CI [-8.0 to 4.5]

5. Secondary Outcome: Number of Participants With Virological Response (Observed, <50 Copies/ml) at Last On-Treatment Visit (Post-Week 96).
Description: Virological response is defined as (observed) plasma viral load less than 50 human immunodeficiency virus-type 1 (HIV-1) ribonucleic acid (RNA) copies per ml at the last on-treatment visit (post-Week 96).
Time Frame: Variable, ranging from 3 months up to maximum 15 months for TMC278 and 12 months for Efavirenz after the 96-week visit
Population: Participants with at least 1 Post-Week 96 visit were included in the analysis.
Measure: Number; unit: Participants
Arm/Group | TMC278 | Efavirenz
Number analyzed (Participants) | 258 | 271
Participants | 245 | 261

6. Secondary Outcome: Number of Participants With Virological Response (Intent-to-Treat - Time to Loss of Virologic Response [TLOVR], <400 Copies/ml) at Week 48
Time Frame: Week 48
Population: The ITT analysis set was considered the primary efficacy analysis set.
Measure: Number; unit: Participants
Arm/Group | TMC278 | Efavirenz
Number analyzed (Participants) | 346 | 344
Participants | 297 | 293

7. Secondary Outcome: Number of Participants With Virological Response (Intent-to-Treat - Time to Loss of Virologic Response [TLOVR], <400 Copies/ml) at Week 96
Time Frame: Week 96
Population: The ITT analysis set was considered the primary efficacy analysis set.
Measure: Number; unit: Participants
Arm/Group | TMC278 | Efavirenz
Number analyzed (Participants) | 346 | 344
Participants | 273 | 278

8. Secondary Outcome: Mean Change From Baseline to Week 48 and Week 96 in Absolute and Relative CD4+ Cell Counts (Using Imputed Data)
Description: Change from baseline in CD4+ cell count was imputed in case of missing values: in case of premature discontinuation, data were imputed with the baseline value after discontinuation (i.e. change=0, Non-Completer [NC] = Failure); otherwise last observation carried forward was applied.
Time Frame: Baseline, Week 48, and Week 96
Population: The ITT analysis set was considered the primary efficacy analysis set.
Measure: Mean (Standard Deviation); unit: cells per microliter
Arm/Group | TMC278 | Efavirenz
Number analyzed (Participants) | 346 | 344
cells per microliter
  Absolute cell count, Week 48 | 195.5 (151.7) | 181.6 (156.9)
  Absolute cell count, Week 96 | 220.7 (167.1) | 226.7 (188.9)
  Relative cell count, Week 48 | 8.6 (5.8) | 8.7 (6.0)
  Relative cell count, Week 96 | 10.1 (7.5) | 10.2 (7.2)

9. Secondary Outcome: Number of Participants With Virologic Failure for the Resistance Determination by Emerging Resistance Associated Mutations: First Available On-Treatment Genotypic Data After Failure
Description: Virologic failure for the resistance determinations was defined as lack of virologic response (never having had 2 consecutive plasma viral load <50 copies/mL) and plasma viral load increase of >=0.5 log 10 copies/mL above nadir (i.e., never suppressed), or confirmed loss of virologic response (2 consecutive plasma viral load >=50 copies/mL after having had 2 consecutive plasma viral load <50 copies/mL; i.e., rebounder), or discontinued with a last observed on-treatment plasma viral load >=50 copies/mL after having had 2 consecutive plasma viral load <50 copies/mL. For this study, treatment-emergent reverse transcriptase (RT) resistance associated mutations (RAMs) occurring in at least 2 virologic failures (for at least one treatment group) for the following lists are presented: i) Extended list of Non-nucleoside reverse transcriptase inhibitor (NNRTI RAMs) ii) IAS-USA list of Nucleoside/tide reverse transcriptase inhibitor (N[t]RTI RAMs).
Time Frame: Week 96
Population: The ITT analysis set was considered the primary efficacy analysis set. Here "N" (Number of Participants Analyzed) signifies number of Participants who were evaluable (had data) for this outcome measure.
Measure: Number; unit: Participants
Arm/Group | TMC278 | Efavirenz
Number analyzed (Participants) | 52 | 18
Participants
  Any RAM from Extended NNRTI RAMs list | 29 | 9
  NNRTI RAM: E138K | 18 | 0
  NNRTI RAM: K101E | 5 | 0
  NNRTI RAM: Y181C | 5 | 0
  NNRTI RAM: V90I | 4 | 0
  NNRTI RAM: V189I | 4 | 0
  NNRTI RAM: H221Y | 4 | 0
  NNRTI RAM: E138Q | 3 | 0
  NNRTI RAM: K103N | 1 | 8
  Any RAM from IAS-USA N(t)RTI RAMs list | 31 | 5
  N(t)RTI RAM: M184I | 24 | 3
  N(t)RTI RAM: M184V | 7 | 3
  N(t)RTI RAM: K065R | 3 | 0
  N(t)RTI RAM: K219E | 3 | 0
  N(t)RTI RAM: Y115F | 2 | 0

ADVERSE EVENTS:
Time Frame: Up to a maximum of 160 weeks for participants in the TMC278 treatment group and up to 147 weeks for participants in the efavirenz treatment group.
Description: Only subjects who had at least one of the TEAEs listed in the Other (non Serious) AE table are included in the Total no. subjects with Non-Serious Adverse Events.
Arm/Group | TMC278 | Efavirenz
Serious Adverse Events (participants affected / at risk) | 40/346 | 43/344
Other Adverse Events (participants affected / at risk) | 231/346 | 268/344
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | TMC278 (N=346) | Efavirenz (N=344)
Abscess limb (Infections and infestations) | 1 | 1
Anogenital warts (Infections and infestations) | 1 | 0
Appendicitis (Infections and infestations) | 1 | 0
Bacterial infection (Infections and infestations) | 1 | 0
Bronchiectasis (Infections and infestations) | 1 | 0
Cellulitis (Infections and infestations) | 2 | 0
Diverticulitis (Infections and infestations) | 1 | 0
Helicobacter gastritis (Infections and infestations) | 1 | 0
Herpes zoster (Infections and infestations) | 1 | 0
Lobar pneumonia (Infections and infestations) | 1 | 0
Neurosyphilis (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 3 | 2
Sepsis (Infections and infestations) | 1 | 0
Syphilis (Infections and infestations) | 1 | 0
Arthritis bacterial (Infections and infestations) | 0 | 1
Bronchitis (Infections and infestations) | 0 | 1
Cerebral toxoplasmosis (Infections and infestations) | 0 | 1
Gastroenteritis (Infections and infestations) | 0 | 1
Streptococcal bacteraemia (Infections and infestations) | 0 | 1
Tuberculous pleurisy (Infections and infestations) | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 0 | 1
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Haemangioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Kaposi's sarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Anal cancer stage 0 (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Burkitt's lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 2
Alcoholism (Psychiatric disorders) | 1 | 0
Depression (Psychiatric disorders) | 2 | 2
Drug dependence (Psychiatric disorders) | 1 | 0
Major depression (Psychiatric disorders) | 1 | 0
Suicide attempt (Psychiatric disorders) | 1 | 0
Bipolar disorder (Psychiatric disorders) | 0 | 1
Homicidal ideation (Psychiatric disorders) | 1 | 1
Haematemesis (Gastrointestinal disorders) | 1 | 0
Peritoneal haemorrhage (Gastrointestinal disorders) | 1 | 0
Anal inflammation (Gastrointestinal disorders) | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 1
Cholecystitis acute (Hepatobiliary disorders) | 1 | 0
Cholelithiasis (Hepatobiliary disorders) | 1 | 1
Cholecystitis (Hepatobiliary disorders) | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Joint swelling (Musculoskeletal and connective tissue disorders) | 1 | 0
Spondylitis (Musculoskeletal and connective tissue disorders) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Calculus ureteric (Renal and urinary disorders) | 1 | 0
Glomerulonephritis membranous (Renal and urinary disorders) | 1 | 0
Chest pain (General disorders) | 1 | 0
Adverse drug reaction (General disorders) | 0 | 1
Pelvic mass (General disorders) | 0 | 1
Pyrexia (General disorders) | 0 | 1
Alcohol poisoning (Injury, poisoning and procedural complications) | 1 | 0
Overdose (Injury, poisoning and procedural complications) | 1 | 0
Drug toxicity (Injury, poisoning and procedural complications) | 0 | 1
Miller fisher syndrome (Nervous system disorders) | 1 | 0
Cerebral ischaemia (Nervous system disorders) | 0 | 1
Cerebrovascular accident (Nervous system disorders) | 0 | 1
Coma (Nervous system disorders) | 0 | 1
Headache (Nervous system disorders) | 1 | 1
Sciatica (Nervous system disorders) | 0 | 1
Cystocele (Reproductive system and breast disorders) | 1 | 0
Uterovaginal prolapse (Reproductive system and breast disorders) | 1 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Erythema (Skin and subcutaneous tissue disorders) | 1 | 0
Rash generalised (Skin and subcutaneous tissue disorders) | 0 | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 1
Atrial flutter (Cardiac disorders) | 0 | 1
Tachycardia (Cardiac disorders) | 0 | 1
Thyroglossal cyst (Congenital, familial and genetic disorders) | 0 | 1
Alanine aminotransferase increased (Investigations) | 0 | 2
Aspartate aminotransferase increased (Investigations) | 0 | 1
Blood alkaline phosphatase increased (Investigations) | 0 | 1
Transaminases increased (Investigations) | 0 | 1
Anorexia (Metabolism and nutrition disorders) | 0 | 1
Bowel preparation (Surgical and medical procedures) | 0 | 1
Drug rehabilitation (Surgical and medical procedures) | 0 | 1
Agranulocytosis (Blood and lymphatic system disorders) | 1 | 0
Splenic lesion (Blood and lymphatic system disorders) | 1 | 0
Coronary artery disease (Cardiac disorders) | 1 | 0
Pyloric stenosis (Congenital, familial and genetic disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0
Anal fissure (Gastrointestinal disorders) | 1 | 0
Liver disorder (Hepatobiliary disorders) | 1 | 0
Anaphylactic reaction (Immune system disorders) | 0 | 1
Bone tuberculosis (Infections and infestations) | 1 | 0
Folliculitis (Infections and infestations) | 0 | 1
Meningococcal sepsis (Infections and infestations) | 0 | 1
Mycobacterium avium complex infection (Infections and infestations) | 1 | 0
Osteomyelitis (Infections and infestations) | 1 | 0
Papilloma viral infection (Infections and infestations) | 0 | 1
Respiratory tract infection (Infections and infestations) | 0 | 1
Tuberculosis (Infections and infestations) | 1 | 0
Ankle fracture (Injury, poisoning and procedural complications) | 1 | 0
Concussion (Injury, poisoning and procedural complications) | 0 | 1
Facial bones fracture (Injury, poisoning and procedural complications) | 0 | 1
Injury (Injury, poisoning and procedural complications) | 1 | 0
Jaw fracture (Injury, poisoning and procedural complications) | 0 | 1
Poisoning (Injury, poisoning and procedural complications) | 1 | 0
Sternal fracture (Injury, poisoning and procedural complications) | 1 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 1
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Anal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Hepatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Hepatic neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Acute psychosis (Psychiatric disorders) | 1 | 0
Panic attack (Psychiatric disorders) | 0 | 1
Psychotic disorder (Psychiatric disorders) | 0 | 2
Suicidal ideation (Psychiatric disorders) | 3 | 1
Asphyxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Circulatory collapse (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | TMC278 (N=346) | Efavirenz (N=344)
Upper respiratory tract infection (Infections and infestations) | 53 | 51
Nasopharyngitis (Infections and infestations) | 45 | 44
Influenza (Infections and infestations) | 37 | 34
Headache (Nervous system disorders) | 50 | 44
Dizziness (Nervous system disorders) | 28 | 91
Somnolence (Nervous system disorders) | 14 | 24
Nausea (Gastrointestinal disorders) | 44 | 38
Diarrhoea (Gastrointestinal disorders) | 51 | 61
Abnormal dreams (Psychiatric disorders) | 29 | 41
Insomnia (Psychiatric disorders) | 36 | 39
Depression (Psychiatric disorders) | 25 | 21
Anxiety (Psychiatric disorders) | 9 | 27
Rash (Skin and subcutaneous tissue disorders) | 26 | 42
Fatigue (General disorders) | 20 | 31
Vomiting (Gastrointestinal disorders) | 15 | 21
Syphilis (Infections and infestations) | 22 | 15
Arthralgia (Musculoskeletal and connective tissue disorders) | 15 | 20
Back pain (Musculoskeletal and connective tissue disorders) | 23 | 24
Cough (Respiratory, thoracic and mediastinal disorders) | 23 | 20
Pruritus (Skin and subcutaneous tissue disorders) | 8 | 18
Hypertension (Vascular disorders) | 21 | 18

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other